CLINICAL TRIAL: NCT00306813
Title: A Multicenter Phase I/II Trial Evaluating the Safety and Efficacy of Lenalidomide (Revlimid, CC-5013) in Combination With Doxorubicin and Dexamethasone (RAD) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Evaluation of Lenalidomide, Doxorubicin and Dexamethasone (RAD) in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSMM VII
Record Dates: First submitted 2006-03-15; First posted 2006-03-24 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2006-03

CONDITIONS: Relapse; Refractory Multiple Myeloma
Keywords: refractory or relapsed multiple myeloma; CC-5013; Revlimid; lenalidomide; RAD
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Lenalidomide

INTERVENTIONS:
Drug: Revlimid

SUMMARY:
This is a multi-center, open label, uncontrolled, non-comparative phase I/II study in patients with refractory or relapsed multiple myeloma who are eligible for second, third, or fourth line therapy. Patients will be enrolled sequentially into four dose cohorts. The feasibility of administrating Revlimid (R) in combination with Doxorubicin and Dexamethasone (AD) and the MTD of the combination will be determined in the phase I part of the study (Part A). When the MTD has been established, the efficacy of the combination will be further evaluated in the phase II part of the study Part B)

DETAILED DESCRIPTION:
Multiple myeloma is an incurable disease that is characterized by the malignant proliferation of plasma cells. It is the second most common hematological malignancy, is invariable fatal. The primary approach for treatment of multiple myeloma is systemic chemotherapy. Conventional chemotherapy with melphalan and prednisone (MP) has increased the survival from 12-17 months to approximately 3 years. But several other studies have shown that combination therapy with addition of other agents such as cyclophosphamide, nitroureas or anthracyclins does not improve the prognosis of patients with multiple myeloma. During the past few years it has been demonstrated that high dose chemotherapy followed by autologous stem cell transplantation can prolong the overall survival of myeloma patients and therefore became the standard of care for younger patients. Since it has been demonstrated that high dose chemotherapy is also well tolerated by the elderly high dose chemotherapy is recommended for patients up to an age of about 70 if there is no relevant comorbidity. Thus, the development of more effective regimens for the teatment of relapsed or refractory myeloma patients is urgently needed. Treatment with corticosteroids alone can induce responses in both primarily resistant and relapsed patients with myeloma. High pulse dexamethasone (40mg daily d1-4, 9-12 and 17-21) showed response rates of 27% in primarily unresponsive patients and 21% in relapsed patients, which were initially responsive. In combination with anthracyclins like in the VAD-regimen (vincristin, adriamycin, dexamethasone)response rates of about 31% were achieved in primary unresponsive patients whereas the response rate was 65% in patients who relapsed, but had previously responded to therapy. Thus, the combination of dexamethasone with anthracyclines and vincristin achieve a certain anti-myeloma activity in relapsed or refractory patients. Nevertheless due to the neurotoxicity, treatment with vincristin of elderly patients is critical and limited. Therefore substitution of vincristine by a less toxic agent with high anti-myeloma activity like the new thalidomide analogues (see below) could reduce toxicity and improve the therapeutic efficacy of anthracycline and dexamethasone containing regimens. Protocol DSMM VII Page 7/52 29.09.2004 Version 1.1 dexamethasone containing regimens. One interesting drug with substantial anti-myeloma activity in patients with relapsed or refractory myeloma is thalidomide. Thalidomide has been demonstrated to induce remissions in about one third of relapsed myeloma patients if given as a single agent therapy. Response rates evaluated in phase-II studies could be improved up to 55% if thalidomide was administered in combination with other drugs such as glucocorticoids. However substantial side effects were observed such as somnolence, constipation and neuropathy. These observations led to development of derivatives of thalidomide in order to reduce toxicity and to improve efficacy. The thalidomide analogues represent a new class of active drugs based on immunmodulatory and direct anti-myeloma effects which have been demonstrated to have a greater potency to inhibit growth of MM and angiogenesis in vitro and in vivo than thalidomide. In a phase I study heavily pretreated patients with relapsed or refractory myeloma were treated with CC-5013 (RevlimidTM, lenalidomide). Revlimid at doses up to 25 mg/day was safe and well tolerated. The dose-limiting toxicity (DLT) was myelosupression at a dose level of 50 mg/day. In contrast to thalidomide treatment with CC- 5013 showed no significant side effects like somnolence, constipation or neuropathy. In addition 29 % of the subjects achieved a > 50% paraprotein reduction, 71% a reduction of > 25%. Preliminary phase II data showed in about 20 % of relapsed myeloma patients a > 50% reduction of paraprotein, a > 25% reduction could be observed in about 50%. No additional toxicity was observed in combination with dexamethasone. Thus, Revlimid as a single agent is well tolerated and has a profound anti-myeloma activity in patients with refractory or relapsed disease. These data suggest that Revlimid combined with chemotherapy could lead to enhanced anti-myeloma effects with acceptable toxicities. The present study will investigate the safety and the efficacy of intermittent dosing of CC-5013 (Revlimid) combined with Dexamethasone and Doxorubicin in the treatment of relapsed or refractory myeloma. Objectives Primary Objectives

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study

1. Understand and voluntarily sign an informed consent form.
2. Age > 18 years at the time of signing the informed consent form.
3. Multiple myeloma with Durie-Salmon stage II or III and considered to have disease progression after at least 1 previous anti-myeloma regimen (examples: induction chemotherapy followed by stem cell collection and high dose chemotherapy and autologous PBSCT; MP; anthracycline-containing regimen > 3 months ago, any other conventional regimen including thalidomide- or bortezomib containing regimens.
4. Subjects must have not have recieved more than 3 previous anti-myeloma regimens and must be relapsed or refractory following at least one regimen of anti-myeloma therapy.
5. No anthracycline-containing regimen (e.g. VAD) within the last 3 months of study.
6. Subjects may have been previously treated with thalidomide or bortezomib.
7. Radiation therapy after start of the protocol will be considered as treatment failure except when given to treat pathological fractures or preexisting osteolytic lesions.
8. Patients must have measurable levels of myeloma paraprotein in serum (>0.5 g/dl) or urine (>0.2 g excreted in a 24-hour collection sample).
9. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
10. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of starting each cycle. Men and WCBP must agree to use adequate contraceptive methods.
11. Must have a 2-d echocardiogram indicating LVEF ≥ 55% within 42 days prior to first dose of study drug.
12. Life extpectancy > 3 months.

Exclusion criteria:

The presence or any of the following will exclude a subject from study enrollment.

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that makes the patient ineligeble for the study. Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias), pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma.
2. Pregnant or lactating females.
3. Heart failure (EF < 55%).
4. Any of the following laboratory abnormalities Absolute neutrophil count (ANC) <1500/mm3 (1x109/L) Platelet count (PLT) <100000/mm3 Serum creatinine> 2.5 mg/dL SGOT and SGPT > 3 x upper limit of normal (ULN) Serum total bilirubin >1.2 mg/dL
5. Prior history of any other malignancies except for adequately treated basal cell, insitu cervical or breast cancer or other for which the patient has been disease free for 5 years.
6. Known hypersensitivity to thalidomide, dexamethasone and/or anthracyline.
7. Prior use of Revlimid.
8. Anthracycline-containing regimen (e.g. VAD) within the last 3 months of study.
9. Any history of thrombembolic events
10. Use of any standard or experimental anti-myeloma drug therapy within 28 days of study enrolment.
11. Major surgery or radiotherapy within 4 weeks of study enrolment.
12. Active infection requiring antibiotic therapy.
13. Subjects who have received > 300 mg/m2 lifetime cumulative dose of doxorubicin alone, or Doxil® alone, or doxorubicin plus Doxil®.
14. History of cardiac disease, with New York Heart Association Class II or greater (See Appendix VII).
15. Known HIV or hepatitis B or C positive.
16. No more than 3 prior anti-myeloma regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2004-09; Study Completion 2008-12

PRIMARY OUTCOMES:
Part A (phase I)
To determine the safety and maximum tolerated dose (MTD) of
Revlimid in combination with Doxorubicin and Dexamethasone
(RAD) administered as a VAD-like regimen in subjects with relapsed or refractory multiple myeloma.
Part B (Phase II):
To determine the efficacy of RAD as treatment for subjects with relapsed or refractory multiple myeloma by estimating the objective response rate (PR, RR and CR).

SECONDARY OUTCOMES:
Secondary objectives of the study are:
Part A plus Part B
To determine the efficacy of RAD as treatment for subjects with relapsed or refractory multiple myeloma by estimating the objective response rate (PR, RR and CR).
To estimate duration of response (PR, RR and CR) and disease control rate (SD, PR and CR).

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bargou, MD, Principal Investigator — Dept. of Internal Medicine II, University of Wuerzburg
Locations (1):
- Dept. of Internal Medicine II, University of Wuerzburg, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Knop S, Gerecke C, Liebisch P, Topp MS, Platzbecker U, Sezer O, Vollmuth C, Falk K, Glasmacher A, Maeder U, Einsele H, Bargou RC. Lenalidomide, adriamycin, and dexamethasone (RAD) in patients with relapsed and refractory multiple myeloma: a report from the German Myeloma Study Group DSMM (Deutsche Studiengruppe Multiples Myelom). Blood. 2009 Apr 30;113(18):4137-43. doi: 10.1182/blood-2008-10-184135. Epub 2009 Jan 30. PMID 19182205